CLINICAL TRIAL: NCT00041340
Title: Phase II Study Of Gleevec (Imatinib Mesylate Formerly Known As(STI571) (NSC #716051) In Patients With Colorectal Cancer Stage IV
Brief Title: Imatinib Mesylate in Treating Patients With Stage IV Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02479; ID01-557; N01CM62202 (NIH); CDR0000069475 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate twice daily. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients with stable disease or better continue therapy until disease progression or 1 year after complete response.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have stage IV colorectal cancer. Imatinib mesylate may interfere with the growth of tumor cells by blocking certain enzymes necessary for cancer cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine response to Gleevec (Imatinib Mesylate) in patients with metastatic colorectal cancer and with c-Kit, Arg, Abl, or PDGF-R expression.

II. To determine the side effects of Imatinib Mesylate in patients with colorectal cancer.

III. To study the biologic effects of Imatinib Mesylate on the c-Kit and PDGF-R system and downstream signaling in metastatic colorectal cancer.

OUTLINE:

Patients receive oral imatinib mesylate twice daily. Treatment continues for 8 weeks in the absence of disease progression or unacceptable toxicity. Patients with stable disease or better continue therapy until disease progression or 1 year after complete response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV colorectal cancer
* Arg, KIT (CD117), or PDGF-R expression (1+ in 20% of cells) in the tumor or microvasculature
* At least one unidimensionally measurable lesion

  * At least 10 mm by spiral CT scan
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* At least 12 weeks
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 2.0 mg/dL
* AST/ALT less than 2.5 times upper limit of normal
* Creatinine no greater than 2.0 mg/mL
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* No other malignancy within the past 3 years except non-melanoma skin cancer or carcinoma in situ of the cervix
* No concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* More than 4 weeks since prior radiotherapy and recovered
* More than 3 weeks since prior surgery (excluding diagnostic biopsy)
* No other concurrent investigational agents
* No concurrent therapeutic doses of anticoagulants (e.g., warfarin)
* No concurrent grapefruit
* No concurrent combination antiretroviral therapy for HIV-positive patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2002-05; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Razelle Kurzrock, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States